CLINICAL TRIAL: NCT07042802
Title: An Open-label, Multicenter Phase Ib/Ⅱ Study to Evaluate the Efficacy and Safety of LBL-024 in Combination With Paclitaxel Injection in Patients With Platinum-resistant Ovarian Cancer
Brief Title: A Phase Ib/Ⅱ Clinical Trial of LBL-024 Combined With Paclitaxel in Patients With Platinum-resistant Ovarian Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanjing Leads Biolabs Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LBL-024-CN006
Record Dates: First submitted 2025-06-17; First posted 2025-06-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Injections; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LBL-024+paclitaxel (Experimental): Experimental group：LBL-024+Paclitaxel.
  LBL-024 and Paclitaxel Intravenous infusion.
  Interventions: Drug: LBL-024 for Injection; Drug: Paclitaxel Injection
- Paclitaxel (Active Comparator): control group： Paclitaxel.
  Paclitaxel Intravenous infusion.
  Interventions: Drug: Paclitaxel Injection

INTERVENTIONS:
Drug: LBL-024 for Injection — LBL-024 Intravenous infusion.
  Other Names: LBL-024
  Arms: LBL-024+paclitaxel
Drug: Paclitaxel Injection — Paclitaxel Intravenous infusion.
  Other Names: Paclitaxel

SUMMARY:
This trial is an open-label, multicenter phase Ib/II clinical study of LBL-024 combination therapy in patients with platinum-resistant ovarian cancer (OC),To evaluate the efficacy and safety of LBL-024 combination therapy in the treatment of advanced recurrent platinum-resistant ovarian cancer (OC) patients.

DETAILED DESCRIPTION:
The trial was divided into two phases.

Stage I (Phase Ib): Single-Arm Safety Lead-In Period. In this stage, a small number of subjects were enrolled first and received LBL-024 combined with paclitaxel treatment, with 21 days as a cycle.Safety, tolerability and preliminary efficacy of combination drugs were assessed by the sponsor and investigators.LBL-024 Dose De-escalation Principle Based on Safety and Tolerability.

Stage II (Phase II) Randomized, Expansion Cohort Study. If safety and tolerability are good, the combined administration extension study will be continued. Subjects were continued to be enrolled in the study. The study was designed as a randomized, open-label, positive-controlled trial.Subjects who met the criteria were randomly assigned to the experimental group and the control group in a ratio of 2: 1.Experimental group (LBL-024 combined with paclitaxel) and Control group (paclitaxel monotherapy).

This study will enroll up to 110 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the trial treatment regimen, visit schedule, laboratory test, and other requirements of the protocol, and voluntarily enroll in the study and sign the written informed consent.
2. At the time of signing the informed consent form, the age was ≥ 18 years old, and the gender was not limited.
3. The Eastern Cooperative Oncology Group's physical status scoring standard (ECOG) is 0~1.
4. The expected survival time is at least 12 weeks.
5. According to the evaluation of RECIST 1.1 （Response Evaluation Criteria in Solid Tumours），the subjects enrolled have at least one measurable lesion.
6. Females of childbearing age are willing to take highly effective contraceptive measures From the signing of the informed consent form to within 6 months after the last administration of the trial drug;Women of childbearing age include pre-menopausal women and women within 2 years after menopause. Women of childbearing age must have a negative pregnancy test within 7 days before the first trial drug is administered.

Exclusion Criteria:

1. The subject is currently participating in any other clinical trial,Or has received or is receiving other investigational agents within 4 weeks prior to the first dose of study drug.
2. Use of immunomodulatory drugs within 2 weeks prior to the first use of study drug.
3. Patients with active infection and currently requiring systemic treatment. active pulmonary tuberculosis (TB), receiving anti-tuberculosis treatment or Received anti-tuberculosis treatment within 6 months before screening.
4. Patients with clinically uncontrollable pleural effusion, pericardial effusion or ascites, and those requiring repeated drainage or medical intervention.
5. The patient has a Medical history of immunodeficiency, including HIV antibody positive.
6. Active hepatitis B or active hepatitis C.
7. Women during pregnancy or lactation.
8. History of mental and/or psychiatric illness (impairing understanding or giving informed consent), drug abuse, alcoholism, or drug addiction.
9. The investigator believes that the subject has other conditions that may affect compliance or are not suitable for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2027-12-25 (Estimated); Study Completion 2028-12-25 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  According to the evaluation criteria of RECIST V1.1 (solid tumour) ,Proportion of subjects achieving complete response (CR) or partial response (PR).It was used to evaluate the efficacy in Phase Ib.
Occurrence of adverse event (AE) and serious adverse event (SAE) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (90 days after drug withdrawal or before the start of new anti-tumor therapy)
  Adverse event (AE) will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0.The safety profile of LBL-024 in combination with paclitaxel will be assessed by monitoring the adverse event (AE) and serious adverse event (SAE) in Phase Ib study.
Progression-free Survival(PFS) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  According to the evaluation criteria of RECIST V1.1 (solid tumour),Time from randomisation to disease progression or death from any cause.It was used to evaluate Time of disease no-progression or Drug resistance in Phase II.

SECONDARY OUTCOMES:
Cmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  Maximum drug concentration in plasma after administration.
Tmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  After administration,Time to reach maximum drug concentration in plasma.
Immunogenicity | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  The immunogenicity is evaluated by the incidence of anti-drug antibodies (ADA) and neutralizing antibodies (if applicable) in subjects.Immunogenicity refers to the performance that can elicit an immune response.
Disease Control Rate(DCR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  Percentage of participants achieving CR, PR, iCR, iPR and stable disease (SD) after treatment.
Duration of Response(DOR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  DOR is defined as the duration from earliest date of disease response (CR、PR 、iCR or iPR) until earliest date of disease progression or death from any cause(if occurring sooner than progression).

CONTACTS AND LOCATIONS:
Overall Officials: lingying wu, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (6):
- China (6):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Tianjin Medical University Cancer Institute &Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No